CLINICAL TRIAL: NCT04810494
Title: Intranasal Lidocaine for Prevention of Postoperative Nausea and Vomiting. A Prospective Double Blind Randomized Controlled Study.
Brief Title: Intranasal Lidocaine for Prevention of Postoperative Nausea and Vomiting.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Change in study team
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Marc Royo, Assistant Professor, Department of Anesthesiology and Perioperative Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00016664
Record Dates: First submitted 2021-03-14; First posted 2021-03-23 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative nausea and vomiting; Intranasal lidocaine
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- test drug (Experimental): 2% Lidocaine
  Interventions: Drug: 2% Lidocaine HCl topical solution
- Placebo (Placebo Comparator): 0.9% Normal Saline
  Interventions: Drug: 0.9% Sodium chloride

INTERVENTIONS:
Drug: 2% Lidocaine HCl topical solution — 0.5mL of 2% Lidocaine will be administered intranasally in each nostril with a mucosal atomization device.
  Arms: test drug
Drug: 0.9% Sodium chloride — 0.5mL of 0.9% Sodium chloride (normal saline) will be administered intranasally in each nostril with a mucosal atomization device.
  Arms: Placebo

SUMMARY:
Postoperative nausea and vomiting (PONV) are common and continue to be persistent problems following general anesthesia. Intranasal lidocaine has been used for the treatment of migraine. The theoretical basis for this effect of intranasal lidocaine on migraine relief is reported to be due to its action on the sodium receptors within the sphenopalatine ganglion. Although there is no reported association between PONV and migraines, injecting lidocaine within the sphenopalatine ganglion has proven to be effective in reducing PONV in endoscopic sinus surgery. The purpose of this study is to investigate the efficacy of intranasal 2% lidocaine in preventing PONV.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is a common complication following general anesthesia.[1] In the absence of prophylaxis, it can occur in greater than one third of the patients undergoing surgery, and the incidence is even higher in patients with predisposing risk factors.[2] Surgical procedures that have been shown to be associated with a high incidence of PONV include breast, gynecologic, abdominal, and thyroid surgeries.[3-5] Although PONV usually resolves with treatment, its occurrence can increase postoperative morbidity, increase hospital cost, and prolong hospital length of stay.[1-6]Despite numerous available prophylactic treatments and proposed strategies, the incidence of PONV continue to be high given its complex pathogenesis.[1]

Lidocaine is a local anesthetic and its intravenous administration has been used as an adjuvant for the treatment of postoperative pain.[7] Intranasal lidocaine has also been used for the treatment of pain, specifically migraine, with significant relief of nausea.[8] The theoretical basis for this effect of intranasal lidocaine on migraine relief is reported to be due to its action on the sodium receptors within the sphenopalatine ganglion.[9] Although there is no reported association between PONV and migraines, injecting lidocaine within the sphenopalatine ganglion has proven to be effective in reducing PONV in patients undergoing endoscopic sinus surgery.[10]

Due to the complex mechanism of PONV, proven benefits of lidocaine on pain and possibly nausea, and previously shown benefit of sphenopalatine block in reducing PONV, we hypothesize that intranasal lidocaine could provide effective prophylaxis for PONV.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age
2. ASA Physical status I-III
3. Ability to provide informed consent
4. Pre-surgical COVID-19 negative test
5. Elective, non-cardiac surgery under general anesthesia including breast surgery, gynecologic surgery, and minimally invasive abdominal surgery

Exclusion Criteria:

1. Local anesthetic allergy
2. Liver diseases
3. Pregnancy
4. Current tobacco use
5. Pre-existing disorders of the gastrointestinal tract
6. Use of anti-emetics within 48 h prior to surgery
7. Chronic use of anti-cholinergic medication or chronic treatment with opioids
8. Any history of nasal pathology (e.g. Nasal ulcer, polyps, and rhinitis)
9. Actual surgical time of <30 min or >180 min
10. Recovery from anesthesia in any location other than PACU
11. History of PONV
12. History of motion sickness
13. Receiving regional blocks for pain management
14. Use of total intravenous anesthesia (TIVA) and/or propofol infusion throughout the case
15. Aprepitant (Emend) administration
16. Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence | up to 1 day
  The incidence of nausea and/or vomiting will be measured by asking the nurse and patient.

SECONDARY OUTCOMES:
Duration of nausea and/or vomiting | up to 1 day
  Duration of nausea and/or vomiting as measured by patient report and physician/nursing observation. This will take place during PACU phase 1.
Rescue treatments | up to 1 day
  Use of pharmacological antiemetics or other rescue treatments for postoperative nausea (PON) or PONV in the PACU (Phase 1). This will include the name of the medications administered, frequency, and doses.
Duration of stay in PACU. | up to 1 day
  Duration (in hours) in PACU phase 1 will be recorded, this is typically up to 4 hours.
Patient satisfaction | At 6 hours after surgery or discharge home, whichever occurs first
  The patients will be asked to grade their satisfaction level as very satisfied, satisfied, dissatisfied, or very dissatisfied)
Intensity | At 6 hours after surgery or discharge home, whichever occurs first
  Intensity will be measured with the validated PONV intensity scale created by Wengritzky et al.[11] This scale ranges from a value of 0 to 50. Clinically important PONV is defined as total score of 50.
Severity | up to 1 day
  Severity of PONV will be measured in PACU phase 1. The severity of PONV will be measured as per the scale described by Eberhart et al.[12] [None (absence of nausea and vomiting), mild (the patient suffered only mild nausea), moderate (the patient suffered 1-2 emetic episodes or moderate or severe nausea without exogenous stimulus and anti-emetics were required), and severe (the patient vomited at least once or experienced nausea at least twice, and anti-emetics were required at least once).

CONTACTS AND LOCATIONS:
Overall Officials: Marc Royo, MD, Principal Investigator — Penn State Health
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Cao X, White PF, Ma H. An update on the management of postoperative nausea and vomiting. J Anesth. 2017 Aug;31(4):617-626. doi: 10.1007/s00540-017-2363-x. Epub 2017 Apr 28. PMID 28455599
- [Background] Obrink E, Jildenstal P, Oddby E, Jakobsson JG. Post-operative nausea and vomiting: update on predicting the probability and ways to minimize its occurrence, with focus on ambulatory surgery. Int J Surg. 2015 Mar;15:100-6. doi: 10.1016/j.ijsu.2015.01.024. Epub 2015 Jan 29. PMID 25638733
- [Background] Tabrizi S, Malhotra V, Turnbull ZA, Goode V. Implementation of Postoperative Nausea and Vomiting Guidelines for Female Adult Patients Undergoing Anesthesia During Gynecologic and Breast Surgery in an Ambulatory Setting. J Perianesth Nurs. 2019 Aug;34(4):851-860. doi: 10.1016/j.jopan.2018.10.006. Epub 2019 Feb 1. PMID 30718165
- [Background] Jeyabalan S, Thampi SM, Karuppusami R, Samuel K. Comparing the efficacy of aprepitant and ondansetron for the prevention of postoperative nausea and vomiting (PONV): A double blinded, randomised control trial in patients undergoing breast and thyroid surgeries. Indian J Anaesth. 2019 Apr;63(4):289-294. doi: 10.4103/ija.IJA_724_18. PMID 31000893
- [Background] Tahir S, Mir AA, Hameed A. Comparison of Palonosetron with Granisetron for Prevention of Postoperative Nausea and Vomiting in Patients Undergoing Laparoscopic Abdominal Surgery. Anesth Essays Res. 2018 Jul-Sep;12(3):636-643. doi: 10.4103/aer.AER_84_18. PMID 30283168
- [Background] Habib AS, Chen YT, Taguchi A, Hu XH, Gan TJ. Postoperative nausea and vomiting following inpatient surgeries in a teaching hospital: a retrospective database analysis. Curr Med Res Opin. 2006 Jun;22(6):1093-9. doi: 10.1185/030079906X104830. PMID 16846542
- [Background] Masic D, Liang E, Long C, Sterk EJ, Barbas B, Rech MA. Intravenous Lidocaine for Acute Pain: A Systematic Review. Pharmacotherapy. 2018 Dec;38(12):1250-1259. doi: 10.1002/phar.2189. Epub 2018 Nov 9. PMID 30303542
- [Background] Vigneault L, Turgeon AF, Cote D, Lauzier F, Zarychanski R, Moore L, McIntyre LA, Nicole PC, Fergusson DA. Perioperative intravenous lidocaine infusion for postoperative pain control: a meta-analysis of randomized controlled trials. Can J Anaesth. 2011 Jan;58(1):22-37. doi: 10.1007/s12630-010-9407-0. PMID 21061107
- [Background] Weibel S, Jelting Y, Pace NL, Helf A, Eberhart LH, Hahnenkamp K, Hollmann MW, Poepping DM, Schnabel A, Kranke P. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery in adults. Cochrane Database Syst Rev. 2018 Jun 4;6(6):CD009642. doi: 10.1002/14651858.CD009642.pub3. PMID 29864216
- [Background] Weibel S, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, Eberhart LH, Poepping DM, Afshari A, Kranke P. Efficacy and safety of intravenous lidocaine for postoperative analgesia and recovery after surgery: a systematic review with trial sequential analysis. Br J Anaesth. 2016 Jun;116(6):770-83. doi: 10.1093/bja/aew101. PMID 27199310
- [Background] Wengritzky R, Mettho T, Myles PS, Burke J, Kakos A. Development and validation of a postoperative nausea and vomiting intensity scale. Br J Anaesth. 2010 Feb;104(2):158-66. doi: 10.1093/bja/aep370. Epub 2009 Dec 26. PMID 20037151
- [Background] Eberhart LH, Seeling W, Ulrich B, Morin AM, Georgieff M. Dimenhydrinate and metoclopramide alone or in combination for prophylaxis of PONV. Can J Anaesth. 2000 Aug;47(8):780-5. doi: 10.1007/BF03019481. PMID 10958095